CLINICAL TRIAL: NCT05252897
Title: Direct Endoscopic Necrosectomy Versus Endoscopic Step-up Approach After Endoscopic Drainage of Walled-off Pancreatic Necrosis (WON)
Brief Title: Timing of Necrosectomy After Endoscopic Drainage of Walled-off Pancreatic Necrosis (WON)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHAN SHANNON MELISSA, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021.465-T
Record Dates: First submitted 2022-02-14; First posted 2022-02-23 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Pancreatic Necrosis
Keywords: walled off pancreatic necrosis; endoscopic drainage; direct endoscopic necrosectomy; endoscopic step up approach
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Intervention Model Description: randomised controlled 2 arm trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic step-up approach (Active Comparator): After endoscopic drainage of WON, patients will be reassessed 72 hours after the procedure. If there is no clinical improvement 72 hours after drain placement, a CECT is performed to check the adequacy of the drainage. Irrigation of the WON via a nasocystic drain or endoscopic irrigation (step 1) is performed in case of inadequate drainage. If a nasocystic drain is inserted, 500ml of normal saline, twice a day will be used to irrigate the WON. If endoscopic irrigation is performed, only irrigation with normal saline without necrosectomy is allowed.
  Patients are again evaluated 72 hours after step 1. In case of improvement, treatment is conservative; otherwise step 2 will be initiated, which is endoscopic necrosectomy. Further endoscopic necrosectomy will be performed until there is clinical improvement.
  Interventions: Procedure: Endoscopic necrosectomy with step up approach
- Direct endoscopic necrosectomy approach (Active Comparator): Patients in the DEN group will undergo an immediate endoscopic necrosectomy after LAMS placement and balloon dilatation. A 10Fr 5cm double pigtail plastic stent will be inserted within the LAMS after necrosectomy. Patients will be assessed in 72 hours after the procedure. If there is no clinical improvement, a CECT is performed to check the adequacy of the drainage. DEN will be repeated in case of inadequate drainage. Patients will be reassessed every 72 hours and DEN repeated until there is clinical improvement. Subsequently, necrosectomy is performed weekly until a reassessment CECT at 3 weeks.
  Interventions: Procedure: Endoscopic necrosectomy with direct approach

INTERVENTIONS:
Procedure: Endoscopic necrosectomy with step up approach — Endoscopic necrosectomy will be performed with a forward-viewing gastroscope into the WON cavity. Debridement of necrotic tissue will be performed with irrigation and/or mechanical removal with endoscopic instruments. For this arm, step up approach will be adopted.
  Arms: Endoscopic step-up approach
Procedure: Endoscopic necrosectomy with direct approach — Endoscopic necrosectomy will be performed with a forward-viewing gastroscope into the WON cavity. Debridement of necrotic tissue will be performed with irrigation and/or mechanical removal with endoscopic instruments. For this arm, the direct approach will be adopted.
  Arms: Direct endoscopic necrosectomy approach

SUMMARY:
Walled-off pancreatic necrosis (WON) is associated with a mortality of 20-30%. The current evidence supports a minimally invasive drainage approach to infected WON. The current suggested approach in international guidelines is the endoscopic step-up approach. However, recent evidence from large national cohorts support the use of direct endoscopic necrosectomy (DEN) at the time of stent placement, resulting in earlier resolution of WON and less number of necrosectomies. This study aims to investigate the clinical outcomes of the DEN versus the step-up approach for necrosectomy after endoscopic drainage of WON.

DETAILED DESCRIPTION:
INTRODUCTION Acute pancreatitis is one of the most common gastrointestinal diseases requiring emergency admissions to the hospital. 10-20% of these patients develop pancreatic necrosis and subsequent walled-off pancreatic necrosis (WON) and is associated with a mortality of 20-30%. Grade 1A evidence exists to support an initial minimally invasive drainage approach to infected WON. However, the optimal approach and timing of necrosectomy remains unaddressed. The current suggested approach in international guidelines is the endoscopic step-up approach. However, recent evidence from large national cohorts support the use of direct endoscopic necrosectomy (DEN) at the time of stent placement, resulting in earlier resolution of WON and less number of necrosectomies.

OBJECTIVE This study aims to investigate the clinical outcomes of the DEN versus the step-up approach for necrosectomy after endoscopic drainage of WON.

HYPOTHESIS The hypothesis is that DEN at the time of LAMS placement improves clinical outcomes after endoscopic drainage of WON as compared to the endoscopic step-up approach.

DESIGN AND SUBJECTS This is a multicentre international randomized controlled trial. Patients with suspected or confirmed infected or symptomatic WON on computed tomography (CT) and who are deemed feasible for endoscopic drainage will be included in the study. Endoscopic drainage with lumen-apposing metal stents (LAMS) will be performed. Patients will be randomised to either the endoscopic step-up approach or direct endoscopic necrosectomy (DEN) approach.

The primary endpoint is a composite of major complications or death within 6 months after randomisation. Secondary endpoints include time to resolution of WON, pancreatic functions, biliary strictures, need for necrosectomy, total number of interventions, length of hospital and ICU stay, recurrence of WON and unplanned readmissions related to WON.

A reduction in cumulative primary endpoint with the DEN approach by 22.4% (32.2% to 9.8%) in comparison to endoscopic step-up approach was assumed. With a 2-sided significance level of 5% and power of 80%, taking into account a 5% drop-out rate, a total of 108 patients was required to demonstrate this effect. Study collaboration has been established with four other international centres. A estimation of 3 years is required to complete study recruitment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥18 years of age) patients
2. Diagnosis of walled-off pancreatic necrosis (WON) based on imaging criteria based on the revised Atlanta classification5
3. Documented history of acute pancreatitis
4. Suspected or confirmed infected WON and/or symptomatic WON causing (i) persistent pancreatic-type pain, and/or ii) gastric outlet or biliary obstruction, and/or (iii) ongoing systemic illness, anorexia, and weight loss, and/or (iv) rapidly enlarging WONs, and/or (v) infected WON*
5. WON identified at contrast-enhanced computed tomography (CECT) and deemed amenable for EUS-guided drainage
6. WON with a solid component >30% and/ or percentage of necrosis >= 30%

Exclusion Criteria:

1. Previous invasive interventions for necrotising pancreatitis
2. An acute flare up of chronic pancreatitis
3. Recurrent acute pancreatitis
4. Indicated for emergency laparotomy (i.e. abdominal compartment syndrome, perforation of a visceral organ, bleeding and bowel ischaemia)
5. Contraindications to endoscopic drainage: previous total gastrectomy, gastric bypass surgery, prior surgery for pancreas-related diseases
6. WON not adherent to the GI wall or not accessible for endoscopic drainage
7. Coagulopathy (INR >1.5), and/or thrombocytopenia (platelets <50,000/mm3)
8. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
A composite of major complications or death within 6 months after randomisation | 6 months
  Major complications include new onset multi-organ failure, multiple organ failure, persistent organ failure, bleeding requiring intervention, perforation of visceral organ requiring intervention, gas embolism

SECONDARY OUTCOMES:
The individual components of the primary endpoint | 6 months
  The individual components include new onset multi-organ failure, multiple organ failure, persistent organ failure, bleeding requiring intervention, perforation of visceral organ requiring intervention, gas embolism
Time to resolution of WOPN | 6 months
  LAMS insertion to LAMS removal
Exocrine pancreatic insufficiency | 6 months
  Exocrine pancreatic insufficiency defined as Oral pancreatic-enzyme supplementation required to treat clinical symptoms of steatorrhea 6 months after randomization; this requirement was not present before onset of acute pancreatitis
Biliary strictures | 6 months
  Presence of biliary strictures on cholangiogram/ CT/ MRI
Total no. of interventions | 6 months
  The total number of interventions including necrosectomy or other surgical/ radiological interventions
Length of hospital | 6 months
  The total length of hospital stay
Recurrence of WOPN | 6 months
  The recurrence of WOPN detected on imaging (CT/ USG/ MRI/ EUS)
Unplanned readmissions related to WOPN | 6 months
  The no. of unplanned readmissions related to WOPN
Endocrine pancreatic insufficiency | 6 months
  Insulin or oral antidiabetic drugs required 6 months after randomization; this requirement was not present before onset of acute pancreatitis
The no. of necrosectomies | 6 months
  The number of necrosectomies required
Total ICU stay | 6 months
  No. of days for ICU stay

CONTACTS AND LOCATIONS:
Locations (9):
- Royal Adelaide Hospital, Adelaide, Australia
- The Chinese University of Hong Kong, Hong Kong, Hong Kong
- India (3):
  - Medanta Institute Of Digestive & Hepatobiliary Sciences, Haryāna
  - Asian Institute of Gastroenterology, Hyderabad
  - Deenanath Mangeshkar Hospital & Research Centre, Pune
- South Korea (2):
  - Asan Medical Centre, Asan
  - SoonChunHyang University School of Medicine, Asan
- Hospital Universitario Rio Hortega, Valladolid, Spain
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No